CLINICAL TRIAL: NCT02727062
Title: Smartphone Pain App for Assessing Oral Mucositis Pain in Patients Receiving Head and Neck Radiation Therapy
Brief Title: Smartphone Pain App for Assessing Oral Mucositis Pain in Patients
Status: Terminated | Type: Observational
Why Stopped: Funding.
Sponsor: Stuart Wong (Other)
Responsible Party: Sponsor-Investigator, Stuart Wong, Professor, Department of Medicine, Division of Hematology/Oncology, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Other Study IDs: PRO0026427
Record Dates: First submitted 2016-03-29; First posted 2016-04-04 (Estimated); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Oral Mucositis
Keywords: head and neck cancer; smartphone application; OM Pain App
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- OM Pain Smartphone Application: This study examines whether the smartphone OM Pain App is a feasible and valid tool to assess pain from radiation-induced oral mucositis.
  Interventions: Device: OM Pain App; Device: Accelerometer

INTERVENTIONS:
Device: OM Pain App — Each study participant will be issued an Android smartphone, or he or she may use his/her own compatible device (whether or not it has an active data service) to which the OM Pain App will be downloaded and installed. Subjects will receive a preprogrammed alarm four times a day from their smartphones prompting them to directly enter OM pain levels on the device. Patients may submit as many pain entries as they wish beyond the four minimum levels.
  Subjects will receive a preprogrammed alarm four times a day from their smartphones prompting them to directly enter OM pain levels on the device. Patients may submit as many pain entries as they wish beyond the four minimum levels.
Device: Accelerometer — Each patient will be issued an accelerometer and will be encouraged to wear it continuously during the study period (weekly during radiation therapy and four weeks following radiation therapy).

SUMMARY:
This research is being done to evaluate whether or not the Oral Mucositis (OM) Pain App (a smartphone application) is a feasible and valid tool to assess pain from radiation sores (also referred to as "mucositis") when treating head and neck cancers with radiation. The mobile app will be designed to help people better understand the pain from the radiation sores.

DETAILED DESCRIPTION:
OVERVIEW: This is a single-arm, observational, supportive care clinical trial for patients with tumors involving the oral cavity, oropharynx, or unknown primary expecting to receive at least a 50 Gy dose of definitive radiation therapy.

OM PAIN APP (DESCRIPTION): The Oral Mucositis (OM) PAIN APP (App) is a smartphone application that was designed to permit patients to key in pain severity, using a visual analog 0-10 scale. The App is programed with an alarm to prompt the patient to record pain severity at prescribed intervals daily and through spontaneous patient input. Data collected on each patient's smartphone can be backed up wirelessly to a central server where the data can be analyzed remotely or data can be viewed on the device. The software is capable of generating a time-weighted measure of pain, total area under the pain cure (AUC), a summary measure that integrates serial assessments of a patient's pain over the duration of the study.

DAILY OBSERVATION: Subjects will receive a preprogrammed alarm four times a day from their smartphones prompting them to directly enter OM pain levels on the device. Patients may submit as many pain entries as they wish beyond the four minimum levels. Data recording will not commence until radiation starts. Because symptoms of mucositis do not commence typically until the third week of radiation therapy, and no sooner than week 2, recordings from week 1 will be used for baseline data. Recording of data will cease four weeks after the end of radiation therapy at which time mucositis symptoms typically start to resolve and pain symptoms substantially abate.

ACCELEROMETER: Each patient will be issued an accelerometer and will be encouraged to wear it continuously during the study period. To help determine whether decline in physical activity is associated with severity of pain, physical activity will be assessed directly with accelerometers (activity monitor). Participants will wear an accelerometer during sleep and waking hours, but not while bathing, starting one week prior to the start radiation therapy. Accelerometer output data will be obtained in 1-minute epochs that will be then summed to provide raw daily average activity units, which will be subsequently divided by 1000 for clarity. Data will by synced weekly by the study coordinator to a computer connected to a central server.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy (including non-squamous cell histologies and unknown primary tumors).
* Patient must be undergoing a course of radiation therapy (RT) (with or without chemotherapy) including oral cavity and/or oropharynx to a dose of at least 50 Gy (SBRT is not allowed).
* Prior definitive course of RT is allowed.
* Physical exam demonstrating no preexisting mucositis.
* Ability to complete the questionnaire.
* No current oral infection or ongoing toxicity from prior radiotherapy.
* Zubrod Score/Eastern Cooperative Oncology Group (ECOG) Performance status < 2.
* Age ≥ 18 years.
* Concurrent enrollment on interventional trial is allowed.
* English-speaking and literate.

Exclusion Criteria:

* Nasopharyngeal cancer
* Paranasal sinus tumors
* Laryngeal cancer
* Pregnant or lactating women are ineligible as treatment involves unforeseeable risks to the participant and to the embryo or fetus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single-arm, clinical trial for patients with tumors involving the oral cavity, oropharynx, or unknown primary.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
The number of subjects who comply with the compulsory four-time daily pain entries. | Week 1 during radiation therapy.
  The study coordinator will download data and check the equipment weekly for proper functioning and compliance. Patients will be interviewed weekly to assure the device is functioning correctly and that data is being recorded.
The number of subjects who comply with the compulsory four-time daily pain entries. | Week 2 during radiation therapy.
  The study coordinator will download data and check the equipment weekly for proper functioning and compliance. Patients will be interviewed weekly to assure the device is functioning correctly and that data is being recorded.
The number of subjects who comply with the compulsory four-time daily pain entries. | Weekly 3 during radiation therapy.
  The study coordinator will download data and check the equipment weekly for proper functioning and compliance. Patients will be interviewed weekly to assure the device is functioning correctly and that data is being recorded.
The number of subjects who comply with the compulsory four-time daily pain entries. | Week 4 during radiation therapy.
  The study coordinator will download data and check the equipment weekly for proper functioning and compliance. Patients will be interviewed weekly to assure the device is functioning correctly and that data is being recorded.
The number of subjects who comply with the compulsory four-time daily pain entries. | Week 5 during radiation therapy.
  The study coordinator will download data and check the equipment weekly for proper functioning and compliance. Patients will be interviewed weekly to assure the device is functioning correctly and that data is being recorded.
The number of subjects who comply with the compulsory four-time daily pain entries. | Week 6 during radiation therapy.
  The study coordinator will download data and check the equipment weekly for proper functioning and compliance. Patients will be interviewed weekly to assure the device is functioning correctly and that data is being recorded.
The number of subjects who comply with the compulsory four-time daily pain entries. | Week 7 during radiation therapy.
  The study coordinator will download data and check the equipment weekly for proper functioning and compliance. Patients will be interviewed weekly to assure the device is functioning correctly and that data is being recorded.
The number of subjects who comply with the compulsory four-time daily pain entries. | Week 8 post-radiation therapy.
  The study coordinator will download data and check the equipment weekly for proper functioning and compliance. Patients will be interviewed weekly to assure the device is functioning correctly and that data is being recorded.
The number of subjects who comply with the compulsory four-time daily pain entries. | Week 9 post-radiation therapy.
  The study coordinator will download data and check the equipment weekly for proper functioning and compliance. Patients will be interviewed weekly to assure the device is functioning correctly and that data is being recorded.
The number of subjects who comply with the compulsory four-time daily pain entries. | Week 10 post-radiation therapy.
  The study coordinator will download data and check the equipment weekly for proper functioning and compliance. Patients will be interviewed weekly to assure the device is functioning correctly and that data is being recorded.
The number of subjects who comply with the compulsory four-time daily pain entries. | Week 11 post-radiation therapy.
  The study coordinator will download data and check the equipment weekly for proper functioning and compliance. Patients will be interviewed weekly to assure the device is functioning correctly and that data is being recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Wong, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No